CLINICAL TRIAL: NCT02877576
Title: Study of Cerebral Mechanisms of Visual Recognition With Single-unit Recordings of Intra-cerebral Neurons in Epileptic Patients
Brief Title: Single Neurons Responses During Visual Recognition in Epileptic Patients
Acronym: REUNIE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-A01951-48
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2020-07

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Epileptic patient (Experimental): micro-electrode recordings interventions: Implantation of mixed intracerebral electrodes Face detection Face individualization
  Interventions: Procedure: Implantation of mixed intracerebral electrodes; Behavioral: Face detection; Behavioral: Face individualization

INTERVENTIONS:
Procedure: Implantation of mixed intracerebral electrodes — 5 macro electrodes with micro electrodes are implanted in internal temporal structures (amygdala, anterior and posterior hippocampus, rhinal cortex, posterior para-hippocampal gyrus).
  Each electrode has 8 microcontacts, each recording the activity of 0 to 3 neurons (activity of 0 to 120 neurons/patient).
Behavioral: Face detection — Visualization of images of 60 unknown faces and 60 objects that are not faces (object, house, scene, animal, plant, word, letter…). Each image is showed for 500 ms and separated from following image by black screen of 1500 ms. In order to keep patient attention on image, patient will be asked to push a button at color change of fixation cross in the centre of image.
Behavioral: Face individualization — Visualization of images of celebrities (persons known by patient), showed randomly. Each image is showed for 500 ms and separated from following image by black screen of 1500 ms. In order to keep patient attention on image, patient will be asked to push a button at color change of fixation cross in the centre of image.
  Several celebrities are showed, with for each the presentation of 60 images different from that celebrity. 1 to 3 celebrities are showed (60 to 180 total images).

SUMMARY:
The purpose is to evaluate specific capacities of face detection of individual neurons by comparison with their capacity of object detection in medial temporal lobe and ventral temporal cortex in epileptic patients.

Secondary purpose is to evaluate specific capacities of detection of known faces of individual neurons by comparison with their capacity of detection of unknown faces in medial temporal lobe and ventral temporal cortex in epileptic patients.

DETAILED DESCRIPTION:
In this interventional study, patients explored with mixed intracerebral electrodes (micro and macro-contacts) will be presented sets of images (objects, unknown faces, famous faces). Spikes and Multi-Unit-Activity will be recorded and analyzed and compared between conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patient with temporal or occipito-temporal drug-resistant partial epilepsy, symptomatic, needing surgical treatment
* Patient having signed informed consent
* Patient affiliated to social security
* Patient having undergone preliminary medical examination

Exclusion Criteria:

* Persons under legal protection or incapable to consent
* Persons deprived of liberty by juridical or administrative decision
* Patient with severe visual disorders of neurological or ophthalmological origin
* Patients with infection risk according to doctor or surgeon
* Women without effective contraception
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Number of action potential (Difference of neuronal activity) generated successively by visual presentation of 60 photography of different unknown faces and 60 different objects | after electrode implantation, up to 12 days
  Activity (number of action potential) is recorded for each neuron before and after visualization of each image.

SECONDARY OUTCOMES:
Number of action potential (Difference of neuronal activity) generated by visual presentation of 60 photography of a known target face (familiar) and 60 photography of unknown faces (non familiar) | after electrode implantation, up to 12 days
  Activity (number of action potential) is recorded for each neuron before and after visualization of each image.

CONTACTS AND LOCATIONS:
Overall Officials: Louis MAILLARD, Pr, Principal Investigator — Service de Neurologie CHRU de Nancy - Hôpital Central
Locations (1):
- Service de Neurologie, Hôpital Central, CHRU de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le Cam S, Jurczynski P, Jonas J, Koessler L, Colnat-Coulbois S, Ranta R. A Bayesian approach for simultaneous spike/LFP separation and spike sorting. J Neural Eng. 2023 Mar 31;20(2). doi: 10.1088/1741-2552/acc210. PMID 36881899